CLINICAL TRIAL: NCT07070180
Title: Analysis of Psychoneuroimmunological Parameters of Health in Specific Population Groups in Slovakia
Acronym: APNIP
Status: Active, not recruiting | Type: Observational
Sponsor: Comenius University (Other)
Collaborators: Slovak Academy of Sciences (Other Government)
Responsible Party: Sponsor
Other Study IDs: APVV-22-0160
Record Dates: First submitted 2025-05-18; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Immunity; Cytokine Levels; Psychological Adaptation; Resilience; Positive Thinking; Sense of Control; Sense of Coherence; Self-control; Problem Solving; Mindfulness; Adverse Childhood Experience; Psychological Distress; Stress; Stress Response; Depression Symptoms; Anxiety Symptoms; Socio-economic Status
Keywords: psychological immunity; biological immunity; psychoneuroimmunology
MeSH Terms: conditions — Self-Control; Fractures, Stress; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Slovak population sample: Adults aged 18 to 50, with the upper age limit set to account for the natural decline in immune function beyond this age. A total of 600 participants were recruited from three regions: 300 from the Bratislava region, 150 from the Banská Bystrica region, and 150 from the Košice region.
- Individuals receiving inpatient treatment for alcohol addiction at the treatment facility: 100 participants aged 18 to 50 years who undergo psychological, epidemiological, and immunological assessments multiple time points - upon admission, during hospitalisation, and at the conclusion of treatment.

SUMMARY:
This study aims to investigate the links between psychological and biological immunity from the perspective of psychology, epidemiology, and immunology in a general population study sample as well as in a specific group of people in treatment for alcohol addiction.

DETAILED DESCRIPTION:
The study will explore the associations between the level of psychological immunity and the current psychological state of the participants, possible links between the level of psychological immunity in adulthood and adverse childhood experiences, and finally, the association between the psychological immunity and biological immunity expressed by the self- assessed perceived immune status and on a molecular level by quantity of cytokines and in a specific subgroup also by natural killer cells. All this will be studied in a sample of general population as well as in a specific group of people in treatment for alcohol addiction that was chosen based on the known adverse immune-related health effects of excessive alcohol consumption.

ELIGIBILITY:
Inclusion Criteria for 'General Slovak Population Sample':

* Age between 18 - 50 years
* Residency in the respective region for at least five years
* Consent to participate in the study

Exclusion Criteria for 'General Slovak Population Sample':

* Individuals younger than 18 or older than 50 years
* Ongoing acute infectious disease on the day of testing
* Eligible individuals who do not provide informed consent

Inclusion Criteria for the sample 'Individuals receiving inpatient treatment for alcohol addiction at the treatment facility':

* Age between 18 - 50 years
* Admission to treatment for alcohol addiction
* Consent to participate in the study, Treatment completion

Exclusion Criteria for the sample 'Individuals receiving inpatient treatment for alcohol addiction at the treatment facility':

* Individuals younger than 18 or older than 50 years
* Eligible individuals who do not provide informed consent
* Drop-out from alcohol addiction treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 'General Slovak Population Sample' will be selected from adult population aged 18-50 years living in Bratislava, Banská Bystrica and Košice regions. Participants were recruited through media promotion of the research. The study group was selected from the registered volunteers based on stratification by age and sex, with equal representation across the age groups 18-30, 31-40, and 41-50 years.
  The sample 'Individuals receiving inpatient treatment for alcohol addiction at the treatment facility' was selected from patients admitted at addiction treatment facility within 48 hours of their admission. The study sample included 100 volunteers aged 18-50 years.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the correlation between psychological immunity, current health status and cytokine levels as indicators of biological immune function. | At the time of study enrollment for Group 1, at the time of admission in treatment and after completion of 3 months of treatment for Group 2
  The psychological instrument will consist of the Psychological immune competence inventory (PICI) to assess the psychological immunity.
  Current health status will be assessed by the epidemiological instrument that will evaluate self-assessed immune status, overall, mental, and physical health, current long-term conditions, social, and economic status. Units of measure for the questionnaires is a score.
  Cytokine secretion by immune cells will be tested using Bio-Plex ProTM Human Cytokine 17- plex assay according to the instructions of the manufacturer. For the analysis the blood plasma will be used. In each sample the following panel of cytokines will be analysed: G- CSF, GM-CSF, IFN-γ, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12 (p70), IL-13, IL-17A, MCP-1 (MCAF), MIP-1β, TNF-α. Cytokine units of measure are picograms per milliliter.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Bražinová, prof., MD, PhD, Principal Investigator — Comenius University, Faculty of Medicine in Bratislava
Locations (3):
- Slovakia (3):
  - Comenius University Bratislava, Faculty of Arts, Bratislava
  - Comenius University, Faculty of Medicine in Bratislava, Bratislava
  - Slovak Academy of Sciences, Institute of Neuroimmunology, Bratislava

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen BL, Farrar WB, Golden-Kreutz DM, Glaser R, Emery CF, Crespin TR, Shapiro CL, Carson WE 3rd. Psychological, behavioral, and immune changes after a psychological intervention: a clinical trial. J Clin Oncol. 2004 Sep 1;22(17):3570-80. doi: 10.1200/JCO.2004.06.030. PMID 15337807
- [Background] Shields GS, Spahr CM, Slavich GM. Psychosocial Interventions and Immune System Function: A Systematic Review and Meta-analysis of Randomized Clinical Trials. JAMA Psychiatry. 2020 Oct 1;77(10):1031-1043. doi: 10.1001/jamapsychiatry.2020.0431. PMID 32492090
- [Background] Brydon L, Walker C, Wawrzyniak A, Whitehead D, Okamura H, Yajima J, Tsuda A, Steptoe A. Synergistic effects of psychological and immune stressors on inflammatory cytokine and sickness responses in humans. Brain Behav Immun. 2009 Feb;23(2):217-24. doi: 10.1016/j.bbi.2008.09.007. Epub 2008 Sep 20. PMID 18835437
- See also: Information about the study published on the website of Comenius Uniiversity in Slovak language — https://uniba.sk/spravodajsky-portal/detail-aktuality/back_to_page/dotazniky/article/analyza-psychoneuroimunologickych-parametrov-zdravia-vo-vybranych-skupinach-slovenskej-populaci/